CLINICAL TRIAL: NCT00832754
Title: Effects of Restricting the Use of AS-AQ Combination Therapy to Malaria Cases Confirmed by a Dipstick Test: A Cluster Randomised Control Trial
Brief Title: Restricting the Use of Artesunate Plus Amodiaquine Combination Therapy to Malaria Cases Confirmed by a Dipstick Test: A Cluster Randomised Control Trial
Acronym: RDT-ACT
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Kintampo Health Research Centre, Ghana (Other)
Collaborators: London School of Hygiene and Tropical Medicine (Other)
Responsible Party: Prof. Daniel Chandramohan, London School of Hygiene and Tropical Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KHRC1
Record Dates: First submitted 2009-01-29; First posted 2009-01-30 (Estimated); Last update posted 2012-12-21 (Estimated); Status verified 2012-12

CONDITIONS: Malaria
Keywords: malaria; rapid diagnostic test; artemisinin; Ghana
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- RDT+ACT group (Experimental): RDT+ACT group (ACT offered to RDT positive cases only)
  Interventions: Device: RDT; Other: Clinical Judgement as basis for treatment of malaria with ACT
- Clinical judgement+ACT group (Active Comparator): Clinical judgement+ACT group (ACT offered to all suspected cases of malaria by clinical judgement)
  Interventions: Device: RDT; Other: Clinical Judgement as basis for treatment of malaria with ACT

INTERVENTIONS:
Device: RDT — Study children attending RDT+ACT HCs with a febrile illness will be tested with an RDT to confirm malaria and treated with ACT only if they have a positive test for malaria parasite. However if there are signs suggestive of other co-morbidities they will be treated with appropriate medicines in addition to AS+AQ.
Other: Clinical Judgement as basis for treatment of malaria with ACT — Study children attending RDT+ACT HCs with a febrile illness will be tested with an RDT to confirm malaria and treated with ACT only if they have a positive test for malaria parasite. However if there are signs suggestive of other co-morbidities they will be treated with appropriate medicines in addition to AS+AQ.

SUMMARY:
Effective use of Rapid Diagnostic Test (RDT) and artemisinin-based combination therapy (ACT) depends on the accuracy and safety of RDT based treatment practices and on factors related to the health delivery system. We propose to study the accuracy and safety of RDT based diagnosis and treatment of febrile illness, health system determinants of effective use of RDTs and the public health outcomes of RDT based ACT for malaria.A cluster randomised trial of RDT based versus clinical judgment based treatment of febrile illness on the incidence of malaria in <48 month old children will be conducted. Health Centres will be randomly allocated to RDT based treatment or clinical judgment based treatment arm and children under 2years of age from the catchment area of each health centre will be followed for 2 years. The cost effectiveness of RDT based approach will be compare with the clinical judgement based treatment.

DETAILED DESCRIPTION:
Two-stage, four component study Stage I - Component A: Accuracy of RDT and the outcome of treatment based on RDT results Primary outcome:What is the sensitivity and specificity of Paracheck cassettes in Ghana to diagnose malaria?

Stage 1 - Component B: delivery system determinants of effective RDT based ACT Primary outcome: What are the delivery system determinants of effective RDT based ACT?

Stage 2 - Component A: effects of restricted use of ACTs based on RDT results: a randomised controlled trial Primary outcome: Incidence of malaria (fever + any level of parasite density) in < 48 month-old children

Stage 2 - component B: Cost effectiveness analysis:

Primary outcome:What is the cost effectiveness of RDT based ACT for treatment of children under 4 years compared with ACT based on clinical judgement?

ELIGIBILITY:
Inclusion Criteria:

* All children aged less than 48mths reporting to health center with suspected malaria

Exclusion Criteria:

* Children having chronic illnesses such as severe malnutrition and heart disease will be excluded from the study.

Max Age: 48 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3063 (Actual)
Dates: Start 2009-03; Primary Completion 2012-08 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Incidence of malaria (fever + any level of parasite density) in < 48 month-old children (Stage 2, Component A) | Three years

SECONDARY OUTCOMES:
Incidence of severe anaemia (Hb <8 g/dl) in < 48 month old children | Three years

CONTACTS AND LOCATIONS:
Overall Officials: Frank E Baiden, Principal Investigator — Kintampo Health Research Center; Jayne Webster, Principal Investigator — London School of Hygiene and Tropical Medicine; Christopher Whitty, Principal Investigator — London School of Hygiene and Tropical Medicine; Seth Owusu-Agyei, Principal Investigator — Kintampo Health Research Center; Daniel Chandramohan, Principal Investigator — London School of Hygiene and Tropical Medicine; Jane Bruce, Principal Investigator — London School of Hygiene and Tropical Medicine
Locations (1):
- Kintampo Health Research Center, Kintampo, BAR, Ghana

REFERENCES:
- [Derived] Tawiah T, Hansen KS, Baiden F, Bruce J, Tivura M, Delimini R, Amengo-Etego S, Chandramohan D, Owusu-Agyei S, Webster J. Cost-Effectiveness Analysis of Test-Based versus Presumptive Treatment of Uncomplicated Malaria in Children under Five Years in an Area of High Transmission in Central Ghana. PLoS One. 2016 Oct 3;11(10):e0164055. doi: 10.1371/journal.pone.0164055. eCollection 2016. PMID 27695130
- [Derived] Baiden F, Bruce J, Webster J, Tivura M, Delmini R, Amengo-Etego S, Owusu-Agyei S, Chandramohan D. Effect of Test-Based versus Presumptive Treatment of Malaria in Under-Five Children in Rural Ghana--A Cluster-Randomised Trial. PLoS One. 2016 Apr 7;11(4):e0152960. doi: 10.1371/journal.pone.0152960. eCollection 2016. PMID 27055275
- [Derived] Baiden F, Webster J, Tivura M, Delimini R, Berko Y, Amenga-Etego S, Agyeman-Budu A, Karikari AB, Bruce J, Owusu-Agyei S, Chandramohan D. Accuracy of rapid tests for malaria and treatment outcomes for malaria and non-malaria cases among under-five children in rural Ghana. PLoS One. 2012;7(4):e34073. doi: 10.1371/journal.pone.0034073. Epub 2012 Apr 13. PMID 22514617